CLINICAL TRIAL: NCT02884518
Title: Predicting Successful Antipsychotic Discontinuation in the First Episode Psychosis by Using Positron Emission Tomography(PET) withPositron Emission Tomography With 3,4-dihydroxy-6-18-fluoro-l-phenylalanine ([18 Fluorine(F)]DOPA)
Brief Title: Predicting Antipsychotic Discontinuation in Psychosis
Acronym: PADP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Euitae Kim, professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: [18F]DOPA PET-1000-1.2
Record Dates: First submitted 2016-08-04; First posted 2016-08-31 (Estimated); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia
Keywords: dopamine receptor occupancy; antipsychotics; positron emission tomography
MeSH Terms: conditions — Schizophrenia | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- patient group (Experimental): The patient group recruits subjects diagnosed with first episode psychosis which occurred within 2 years and having been treated with antipsychotics for 1 year. Subjects in the patient group will receive a reduced intake of antipsychotics by 25% after each week of the four-week period in which they will also undergo PET imaging at the baseline, 7 week, and 8 week marks to detect the correlation between the capacity. And patient group should complete clinical scales at 0, 2, 4, 6, and 8 week.
  Interventions: Device: PET; Behavioral: clinical scale
- healthy control group (Other): Screening tests for healthy volunteers included physical examination, vital signs, laboratory will test (hematology, blood chemistry, and urinalysis), and a 12-lead electrocardiograms. A psychiatric interview with the Structured Clinical Interview for text revision of the Diagnostic and Statistical Manual of Mental Disorders -IV(DSM-IV-TR) Axis I disorders, Research Version, Nonpatient Edition (SCID-I/NP) (First et al. 2002) will be conducted. Subjects with any medically significant abnormality on investigations and/or psychiatric disease will be excluded. Also, healthy control group will take a PET scan at 0, 2, 4, 6, and 8 week and clinical scales at baseline.
  Interventions: Device: PET; Behavioral: clinical scale

INTERVENTIONS:
Device: PET — Subjects in the patient group will receive a reduced intake of antipsychotics by 25% after each week of the four-week period in which they and healthy controls will also undergo PET imaging at the baseline, 7 week, and 8 week marks to detect the correlation between the capacity of presynaptic dopamine and relapse in the patients discontinuing treatment.
Behavioral: clinical scale — Healthy controls should complete clinical scales at baseline. Patient group should complete clinical scales at 0, 2, 4, 6, and 8 week.

SUMMARY:
The purpose of this study is to determine whether dopamine synthesis capacity by using [18 fluorine(F)]-DOPA PET for patients with schizophrenia in the maintenance phase can predict treatment discontinuation.

DETAILED DESCRIPTION:
There are two groups: the healthy control group (n=12) and the patient group (n=26). The patient group recruits subjects diagnosed with first episode psychosis which occurred within 2 years and having been treated with antipsychotics for 1 year. Participants will complete clinical scales and undergo PET scans. Subjects in the patient group will receive a reduced intake of antipsychotics by 25% after each week of the four-week period in which they will also undergo PET imaging at the baseline, 7 week, and 8 week marks to detect the correlation between the capacity of presynaptic dopamine and relapse in the patients discontinuing treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient group

1. Patients who met DSM-IV criteria for schizophrenia, schizoaffective disorder, and schizophreniform disorder
2. patients diagnosed with first episode psychosis which occurred within 2 years and having been treated with antipsychotics for at least 1 year.
3. Patients who have maintained in the stable state for 3 months without medication change at the baseline.

2. Healthy control group

* Healthy controls has no Axis I disorder and do not report any past event of neurological or psychiatric illness assessed by the Structured Clinical Interview for DSM Disorders

Exclusion Criteria:

1. Participants should not have any neurological illness such as head trauma, seizure and meningitis.
2. Participants should not be diagnosed as Mental retardation(IQ<70)
3. Participants should not have severe personality disorder, substance abuse or dependence (except for nicotine abuse and dependence) and severe medical conditions.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Ki(cer) of 3,4-dihydroxy-6-18-fluoro-l-phenylalanine ([18 fluorine(F)]DOPA PET) | Change from Baseline Ki(cer) of [18 fluorine(F)]DOPA PET at 7 weeks and at 8 weeks
  Subjects in the patient group will receive a reduced intake of antipsychotics by 25% after each week of the six-week period in which they will also undergo PET imaging at the baseline and six-week marks to detect the correlation between the capacity of presynaptic dopamine and relapse in the patients discontinuing treatment.

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale(PANSS)Scale | at 0, 2, 4, 6, and 8 wk
  Psychotic symptoms will be assessed by using PANSS at 0, 2, 4, 6, and 8 wk
Brief Psychiatric Rating Scale(BPRS) | at 0, 2, 4, 6, and 8 wk
  Psychotic symptoms will be assessed by using BPRS at 0, 2, 4, 6, and 8 wk
Young Mania Rating Scale(YMRS) | at 0, 2, 4, 6 and 8 wk
  Mood symptoms will be assessed by using YMRS at 0, 2, 4, 6 and 8 wk
Hamilton Depression Rating Scale(HAM-D) | at 0, 2, 4, 6 and 8 wk
  Mood symptoms will be assessed by using HAM-D at 0, 2, 4, 6 and 8 wk
Columbia Suicide Severity Rating Scale(C-SSR) | at 0, 2, 4, 6, and 8 wk
  Suicide risk will be assessed by using C-SSR at 0, 2, 4, 6, and 8 wk
Quality of Life Scale(QoL) | at 0 , 4 and 8 wk
  QoL will be assessed at 0 , 4 and 8 wk
Adverse effects | at 0 and 4 wk
  Adverse effects will be assessed by using side effect rating scale at 0 and 4 wk
Kv-Subjective Well-Being Under Neuroleptics Scale(SWN)-K | at 0, 4 and 8 wk
  Dysphoria will be assessed by using Kv-SWN-K at 0, 4 and 8 wk

CONTACTS AND LOCATIONS:
Overall Officials: Euitae Kim, Ph. D., Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided